CLINICAL TRIAL: NCT03583801
Title: Aromatherapy and Peri Operative Anxiety : Assessment in Ambulatory Elective Upper Limb Surgery Under Loco-regional Anesthesia, a Randomized Controlled Study
Brief Title: Assessment of the Aromatherapy to Alleviate Peri Operative Anxiety in Ambulatory Elective Upper Limb Surgery Under Loco-regional Anesthesia
Acronym: AROMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017_58; 2018-A00642-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Anxiety
Keywords: Perioperative Anxiety; Aromatherapy; Surgery; Loco-regional Anesthesia; Ambulatory
MeSH Terms: conditions — Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aromatherapy group (Experimental): The patient has to choose an essential oil among the 3 proposed :
  * sweet orange (Citrus sinensis L. Persoon)
  * fine lavender (Lavandula angustifolia P. Miller)
  * little seed from the mandarin tree (Citrus reticulata blanco)
  Interventions: Other: Olfactory aromatherapy
- without aromatherapy (Placebo Comparator)
  Interventions: Other: without aromatherapy

INTERVENTIONS:
Other: Olfactory aromatherapy — 2 drops of the essential oil choosed by the patient are applied on a compress placed next to his head from his arrival in the recovery room to his leaving from the operating theatre. The method of administration is the respiratory tract..
  Other Names: Inhalation of essential oils
  Arms: aromatherapy group
Other: without aromatherapy — no intervention
  Arms: without aromatherapy

SUMMARY:
AROMA study is a randomised controlled parallel-group single-site study. Patients randomized in the experimental group benefit from the aromatherapy at their arrival in the operating theatre in the recovery room. 2 drops of essential oils are applied on a compress placed next to the head of the patient. This compress is kept until the patient is leaving the operating theatre. Patients randomized in the control group don't benefit from the aromatherapy. The anxiety evolution is measured in both groups with the Amsterdam Preoperative Anxiety and Information Scale (APAIS). The hypothesis is that aromatherapy alleviate peri operative anxiety during an ambulatory elective upper limb surgery under loco-regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in Hospital Centre for an ambulatory elective upper limb " fast track " surgery
* Patient with loco-regional anesthesia
* Patient categorized 3 or less according to the American Society of Anesthesiologists (ASA) score
* The patient must have given his written consent to participate in the study
* Patient - insured under the French social security system
* Patient prepared to comply with all the terms of the study and its length

Exclusion Criteria:

* Epileptic patients
* Asthmatic patients
* Patients with cognitive disorders ( Mini Mental Status below 15)
* Psychiatric disorders : current depression or bipolar disease or anxiety disorders or psychotic disorders according to DSM-V classification
* American Society of Anesthesiologists score strictly superior to 3
* Preoperative chronic pain : neuropathic pain, fibromyalgia, polyarthritis
* Pregnant or breastfeeding woman
* Patient unable to receive an informed consent and to comply with all the terms of the study
* Patient without any social insurance
* Refusal to sign the consent
* Patient under legal protection
* Patient in emergency (unstable clinical state)
* Patient unable to read or write french
* Patient enrolled in an other clinical trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Amsterdam Preoperative Anxiety and Information Scale (APAIS) score variation | Between time T0 (arrival in the operating room in the recovery room) and time T1 (10 minutes after T0, before loco-regional anesthesia), an average 10 minutes

SECONDARY OUTCOMES:
Anxiety Visual Analogic Scale change after the arrival in the operating room | at baseline and an average at 10 minutes,at 35 minutes, at 70 minutes and at 3 hours after arriving in operating room
Satisfaction Visual analogic Scale change after the arrival in the operating theater. | at baseline and an average ,at 35 minutes, at 70 minutes and at 3 hours after arriving in operating room
Comfort Visual analogic Scale variation change after the arrival in the operating theater. | at baseline and an average at 35 minutes, at 70 minutes and at 3 hours after arriving in operating room
Percentage of patients needing a perioperative drug-induced sedation. | at baseline and an average ,at 35 minutes, at 70 minutes and at 3 hours after arriving in operating room

CONTACTS AND LOCATIONS:
Overall Officials: Cécile RIVOAL, Principal Investigator — University Hospital, Lille
Locations (1):
- Centre hospitalier, Valenciennes, France